CLINICAL TRIAL: NCT06724718
Title: Diagnosis of Atrial Fibrillation in Postoperative Thoracic Surgery Using a Smartwatch
Acronym: THO-FA-WATCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Clinique Victor Pauchet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2023_843_0139
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Atrial Fibrillation; Thoracic Surgery; Smartwatches; Rhythm Monitoring; Cardiovascular Prognosis; Asymptomatic Atrial Fibrillation; Randomized Trial
Keywords: Postoperative atrial fibrillation; thoracic surgery; smartwatches; rhythm monitoring; cardiovascular prognosis; asymptomatic atrial fibrillation; randomized trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smartwatch group (Experimental): Experimental intervention using smartwatches for rhythm monitoring.
  Interventions: Other: smartwatch; Other: ECG
- Control group (Active Comparator): Standard care without smartwatch monitoring
  Interventions: Other: ECG

INTERVENTIONS:
Other: smartwatch — Patients in the smartwatch group will undergo rhythm monitoring with a smartwatch
  Arms: Smartwatch group
Other: ECG — Detected POAF episodes will be confirmed via a 12-lead ECG

SUMMARY:
Postoperative atrial fibrillation (POAF) occurs in approximately 20% of patients following thoracic surgery. Early diagnosis is essential to prevent complications such as heart failure, stroke, myocardial infarction, and increased mortality. Smartwatches equipped with single-lead ECG capabilities and algorithms to detect asymptomatic atrial fibrillation (AF) offer a potential solution. This study aims to evaluate the effectiveness of smartwatches in detecting POAF compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years old).
* Patients undergoing major thoracic surgery with one-lung ventilation within the past 48 hours.
* Scheduled pneumonectomy or lobectomy.
* Admission to a conventional surgical unit postoperatively.
* Ability to perform single-lead ECG using a smartwatch.
* Coverage under a social security system.
* Signed informed consent

Exclusion Criteria:

* History of atrial fibrillation.
* Requirement for telemetry for AV block or tachyarrhythmias (>140 bpm).
* Dependency on a pacemaker.
* Participation in another interventional clinical trial affecting POAF incidence.
* Mediastinal, pleural, or chest wall surgery.
* Reoperations or surgeries performed more than 48 hours prior.
* Pregnant women.
* Patients under guardians or similar legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of POAF | at day 7
  the incidence of POAF within seven days after scheduled thoracic surgery.

SECONDARY OUTCOMES:
Rate of asymptomatic POAF | at day 7
  Rate of asymptomatic POAF, evaluated using the EHRA symptom score
Cardiovascular prognosis | at day 3
  Cardiovascular prognosis assessed through a composite outcome (MACE)
Cardiovascular prognosis | at 6 months
  Cardiovascular prognosis assessed through a composite outcome (MACE)
Feasibility of rhythm monitoring with a smartwatch | at day 7
  Feasibility of rhythm monitoring with a smartwatch, measured by device usage time and the proportion of successful single-lead ECGs performed.
Recurrence of AF | at 3 months
  Recurrence of AF
Recurrence of AF | at 6 months
  Recurrence of AF
management of AF | at 3 months
  management of AF
management of AF | at 6 months
  management of AF

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Huette, MD, Principal Investigator — Centre Hospitalier Amiens
Locations (1):
- Centre hospitalier Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huette P, Beyls C, Diouf M, Ibrahima A, Haye G, Guilbart M, Lefebvre T, Bayart G, Lhotellier F, Radji M, Walczak KA, Caboche M, De Dominicis F, Georges O, Berna P, Merlusca G, Hermida A, Traulle S, Dupont H, Mahjoub Y, Abou-Arab O; THOFAWATCH Study Group. Study protocol: diagnosis of atrial fibrillation in postoperative thoracic surgery using a smartwatch, an open-label randomised controlled study (THOFAWATCH trial). BMJ Open. 2025 Apr 9;15(4):e097765. doi: 10.1136/bmjopen-2024-097765. PMID 40204329